CLINICAL TRIAL: NCT00146263
Title: The Effect of Computerized Cognitive Training on Neuropsychological Measures of Cognitive Function in the Elderly
Brief Title: Computerized Cognitive Training in the Elderly
Acronym: CogTrain
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Difficulty in enrolling subjects in the proposed crossover study design
Sponsor: Beersheva Mental Health Center (Other Government)
Responsible Party: Principal Investigator, Tzvi Dwolatzky, Principal Investigator, Beersheva Mental Health Center
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: BMHC-4018CTIL
Record Dates: First submitted 2005-09-04; First posted 2005-09-07 (Estimated); Last update posted 2020-02-27 (Actual); Status verified 2020-02

CONDITIONS: Dementia
Keywords: mild cognitive impairment; dementia; Alzheimer's Disease; cognitive training
MeSH Terms: conditions — Dementia; Cognitive Dysfunction; Alzheimer Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Savyon (Active Comparator): Computerized cognitive training using the Savyon software
  Interventions: Behavioral: Savyon
- Control (Placebo Comparator): Usual activity
  Interventions: Behavioral: Control

INTERVENTIONS:
Behavioral: Savyon — Computerized cognitive training
  Arms: Savyon
Behavioral: Control — Usual activity
  Arms: Control

SUMMARY:
Background:

The aging of the population has lead to a significant increase in the number of older people suffering from cognitive impairment and dementia. The present lack of effective drug therapy for these conditions makes it imperative to investigate other potential therapeutic interventions.

Cognitive training has been described as possibly useful in improving cognitive function in elderly subjects with mild impairment and early dementia. However, there have been few well-designed studies to date and the results are equivocal. Most studies have relied on the use of paper-based neuropsychological assessment instruments with limited accuracy and reproducibility. The investigators have developed a validated computerized neuropsychological assessment battery with increased test-retest reliability.

The purpose of this study is to assess the efficacy of a computerized training program on cognitive function in older persons with normal cognition, mild cognitive impairment, and early dementia.

Description:

A randomized prospective AB/BA crossover study.

Methods:

Eligible males and females aged 60 years and older following initial computerized neuropsychological assessment will be randomized to receive either a 12-session computerized cognitive training program, or no treatment. Repeat neuropsychological assessment will be followed by a 4-week no treatment phase, reassessment and crossover phase.

DETAILED DESCRIPTION:
Background

In recent years there has been an increase in the elderly population. This fact has led to a significant number of people suffering from diseases which are associated with old age, amongst which is dementia.

The medical treatment of dementia is limited in its effectiveness and thus it is important to investigate other methods of therapy. One of the possible options to preserve the cognitive function is to apply cognitive exercise. If these exercises can improve cognitive expertise, it would open new vistas of treatment for dementia patients.

From a few research projects that have taken place on the subject, it has not been proved that cognitive exercising has been of use to patients suffering from mild dementia mainly because of methodological restraints. Thus it is necessary to undertake controlled random research on the subject.

The assessment of the cognitive state and the change in its status demands sensitive measurements. Objective and accurate computerized neuro-physiological testing like "Mindstream ®" and computer hardware are readably available. This technique enhances motivation and encourages participation.

Purpose of the work:

To evaluate the influence of computerized cognitive exercise on the cognitive function of the elderly suffering from mild dementia.

Methods:

IA randomized controlled study using a crossover AB/BA design will be performed. The intervention group will participate in a 12-session twice weekly intervention using the "Savyon" computerized cognitive training program (developed by the Melabev organization Jerusalem), which includes memory, language, arithmetic exercises and puzzles matching colors and shapes. The control group will continue with usual activities with no additional cognitive stimulation. Following a 4-week "washout" phase the groups will be switched in an AB/BA crossover design. A total of 150 subjects with mild cognitive impairment or early dementia will be included. Primary outcome measure will be the Mindstreams® (NeuroTrax Corp., N.Y.) computerized cognitive assessment battery performed initially, at 12 weeks, 16 weeks, 28 weeks.

For each Mindstreams ® index, the differences were compared the testing within each group utilizing "Wilcoxon Signed Ranks test" and between the groups utilizing "Mann-Whitney U test".

ELIGIBILITY:
Inclusion Criteria:

* Age: above 60 years old

Exclusion Criteria:

* Visual impairment
* Educational inability to perform training

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2005-09; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
Computerized cognitive assessment using the Mindstreams battery | 12 weeks
  Changes in cognitive function including memory, executive function, visual spatial and attention.

CONTACTS AND LOCATIONS:
Overall Officials: Tzvi Dwolatzky, MD, Principal Investigator — Ben-Gurion University of the Negev
Locations (1):
- Beersheva Mental Health Center, Beersheva, Israel

IPD SHARING:
Plan to Share IPD: No